CLINICAL TRIAL: NCT05921370
Title: Effect of Perioperative Silodosin on Ureteric Dilatation in Retrograde Intrarenal Surgery
Brief Title: Silodosin in Retrograde Intrarenal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS 231/2023
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis | interventions — silodosin

STUDY DESIGN:
Intervention Model Description: This prospective study will be conducted in patients prepared for RIRS presented to Ain Shams University Hospital.
  Group A (the study group): Patients will receive silodosin 8 mg one tablet per day for 7 days Group B (the control group): Patients will receive Placebo for 7 days before their scheduled retrograde intrarenal surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silodosin group (the intervention group) (Experimental): Patients will receive silodosin 8 mg one tablet per day for 7 days before their scheduled retrograde intrarenal surgery.
  Interventions: Drug: Silodosin 8 mg
- Placebo group (the control group) (Placebo Comparator): Patients will receive Placebo for 7 days before their scheduled retrograde intrarenal surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin 8 mg — This prospective study will be conducted on patients prepared for Retrograde intrarenal surgery presented to Ain Shams University Hospital. Patients will be randomized with 1:1 ratio into 2 equal groups.
  Group A (the study group): Patients will receive silodosin 8 mg one tablet per day for 7 days before their scheduled retrograde intrarenal surgery.
  silodosin is an alpha blocker which act to dilate the ureter to facilitate access sheath placement
  Arms: Silodosin group (the intervention group)
Drug: Placebo — This prospective study will be conducted on patients prepared for Retrograde intrarenal surgery presented to Ain Shams University Hospital. Patients will be randomized with 1:1 ratio into 2 equal groups.
  Group A (the study group): Patients will receive silodosin 8 mg one tablet per day for 7 days before their scheduled retrograde intrarenal surgery.
  Group B (the control group): Patients will receive Placebo for 7 days before their scheduled retrograde intrarenal surgery.
  Arms: Placebo group (the control group)

SUMMARY:
Selective alpha-blockers have been used for the treatment of ureteric stones as medical expulsive therapy (MET). Recently they have been successfully used in passive ureteric dilatation before semirigid ureteroscopy. This study enables us to know the role of silodosin in ureteric dilatation to facilitate ureteral access sheath placement in Retrograde Intrarenal Surgery with flexible ureteroscopy.

DETAILED DESCRIPTION:
The ureteral access sheaths (UAS) used during Retrograde Intrarenal Surgery (RIRS) were produced for easy access to the upper urinary tract. The main advantages of UAS are providing repetitive access to the ureteral and collecting duct system, decreasing intrarenal pressure, preventing bleeding-related distortion of vision by the acceleration of liquid flow, and eventually contributing toward the protection of the flexible device.

Nevertheless, there might be certain challenges during UAS placement. There are also risks, such as ureteral injury and the occurrence of ureteral stricture in the long term. However, considering the benefit/risk balance, RIRS is routinely performed in many clinics because of the ease provided by UAS.

Some problems might occur during the placement of UAS whose diameters vary between 9.5 and 14 Fr. In cases where UAS cannot be placed, manipulations can be used, such as ureteral balloon dilatation, providing access through a rigid ureteroscope with a guide wire, or dilatation with the inner sheath of the UAS, which may vary depending on the amount of personal experience. Despite such manipulations, if UAS placement is still unsuccessful, it is always more logical to place a double-J stent, enables passive dilatation, and postpone RIRS until the second operation.

This study will examine whether intramural ureteral resistance can be reduced or not and whether UAS placement can be facilitated using silodosin or not.

ELIGIBILITY:
Inclusion Criteria:

* Both sex.
* Age >18 yrs old.
* Upper ureteric stones or renal stones < 2 cm.
* Patients with normal renal anatomy.
* No history of infectious or inflammatory renal condition.

Exclusion Criteria:

* • < 18 years old.

  * Multiple or bilateral stones.
  * Pregnant women.
  * Ureteric strictures.
  * Urinary tract infection.
  * Coagulopathy and uncorrected bleeding disorders.
  * Refusal of the surgery and requiring stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
ureteric access sheath placement | intraoperative immediate diagnosis, at the beginning of surgery.
  to assess the success of ureteric access sheath placement as follows:
  1. Direct assessment: A. Success of ureteric access sheath insertion without ureteric dilatation. B. Success of ureteric access sheath insertion with ureteric dilatation. C. Failed ureteric access sheath insertion.

SECONDARY OUTCOMES:
operative time | intraoperative diagnosis during the surgery from beginning of the surgery till the end of the procedure
  time of the procedure will be recorded from the beginning of the diagnostic cystoscopy till placement of the flexible ureteroscopy
Perioperative complication | till 7 days postoperative
  regarding of both intraoperative complications in the form of ureteric mucosal tear, ureteric avulsion, residual stones, postoperative pain, dysuria, hematuria, and fever
Cost analysis | 1 day post operative
  evaluation of the cost in both arms by comparing the price for the medication for 7 days on one arm. and the cost of the supplies needed intraoperative for ureteric dilatation or the need for another surgical session

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided